CLINICAL TRIAL: NCT06680102
Title: The Effectiveness of Weizmannia Coagulans BC99 in Alleviating Allergic Rhinitis in Adults and Its Impact on the Gut Microbiota.
Brief Title: Probiotic Ameliorates Adult Allergic Rhinitis and Modulates Gut Microbiota
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: WK2024010
Record Dates: First submitted 2024-11-04; First posted 2024-11-08 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2024-09

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Probiotic soft candies containing Weizmannia coagulans BC99, 10 billion CFU per piece, to be chewed directly, 2 pieces daily.
  Storage method: Keep away from light, seal tightly, and store in a cool, dry place.
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Gummies without Weizmannia coagulans BC99, to be chewed directly, 2 pieces per day.
  Storage method: Keep away from light, seal tightly, and store in a cool, dry place.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The experimental phase of this study lasts for 8 weeks, with each patient making three visits at weeks 1, 4, and 8.
  Arms: Probiotic Group
Dietary Supplement: Maltodextrin — The experimental phase of this study lasts for 8 weeks, with each patient making three visits at weeks 1, 4, and 8.
  Arms: Placebo Group

SUMMARY:
Assessing the clinical efficacy of weizmannia coagulans BC99 in alleviating allergic rhinitis symptoms, improving gut microbiota, and reducing adverse reactions in patients.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily and in writing, sign an informed consent form agreeing to participate in this study;
2. Able to complete the study as required by the trial protocol;
3. Age between 18 and 65 years old;
4. Meet the diagnostic criteria for allergic rhinitis established in the "Chinese Guidelines for the Diagnosis and Treatment of Allergic Rhinitis (2022 Revised Edition)";
5. Symptoms: Presence of two or more symptoms such as sneezing, watery rhinorrhea, nasal itching, and nasal congestion, with daily symptoms lasting or accumulating for more than 1 hour, which may be accompanied by eye itching, tearing, and redness of the eyes and other ocular symptoms;
6. Signs: Pale and edematous nasal mucosa, which may be accompanied by watery secretions.

Exclusion Criteria:

1. Use of drugs affecting the gut microbiota (including antimicrobial agents, probiotics, intestinal mucosal protective agents, traditional Chinese patent medicines, etc.) for more than 1 week within 1 month prior to screening;
2. Patients with coexisting pulmonary tuberculosis;
3. Patients with coexisting allergic asthma;
4. Patients with nasal polyps or severe nasal septum deviation;
5. Patients with severe systemic diseases or malignant tumors;
6. Individuals with congenital genetic diseases or congenital immunodeficiency diseases;
7. Regular use of probiotics or prebiotics within 6 months prior to the screening period;
8. Patients with severe gastrointestinal diseases (including severe diarrhea, inflammatory bowel diseases, etc.);
9. Individuals with metabolic syndrome (including obesity, dyslipidemia, hypertension, diabetes, etc.);
10. Patients with sinusitis, otitis media, or respiratory tract infections;
11. Individuals allergic to any components of the probiotics used in this trial;
12. Pregnant or lactating women or those planning to conceive in the near future;
13. Those who discontinue the test sample or take other medications midway, making it impossible to determine efficacy or with incomplete data;
14. Recent use of products similar to the test function, affecting the judgment of the results;
15. Participants who cannot participate in the trial due to their own reasons;
16. Other participants deemed ineligible by the researcher.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2024-12-25 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
Improvement of rhinitis symptoms in participants | 8 weeks
  Improvement in Nasal symptoms was assessed using the Total Nasal Symptom Score(TNSS), which included four common nasal symptoms: itchiness, nasal congestion, sneezing, and runny nose. The four symptoms were scored using a "four-point scale", that is, according to the severity of each symptom from 0 to 3 points, that is, the higher the score, the more severe the symptoms, and the total score of the entire TNSS score is the sum of the four symptom scores, which ranges from 0 to 12 points.

SECONDARY OUTCOMES:
16S rRNA sequencing was used to evaluate the changes of intestinal flora before and after the intervention | 8 weeks
  Changes in subjects' fecal microbiota, including abundance and proportion of beneficial bacteria, were assessed by 16S rRNA sequencing before and after probiotic intervention.
Effect of probiotic intervention on immunoglobulin in subjects | 8 weeks
  The changes of Immunoglobulin A and Immunoglobulin E before and after intervention were detected by ELISA.
Impact on Serum Inflammatory Cytokines | 8 weeks
  Levels of IL-4, IL-5, IL-10, IL-13.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Food and Bioengineering, Henan University of Science and Technology, Luoyang, Henan, China

REFERENCES:
- [Derived] Li X, Han Z, Wu K, Lin B, Azeem S, Jiang Y, Dong Y, Gai Z, Fang S, Wu Y, Gu S. Weizmannia coagulans BC99 regulates oxidative stress and serum metabolic pathways to improve allergic rhinitis: a randomized, double-blind, placebo-controlled trial. Front Immunol. 2025 Oct 24;16:1654724. doi: 10.3389/fimmu.2025.1654724. eCollection 2025. PMID 41208993